CLINICAL TRIAL: NCT03899402
Title: Triple Therapy for Type 1 Diabetes With Insulin, Semaglutide, and Dapagliflozin
Brief Title: Triple Therapy in T1DM
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: University of Glasgow (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, paresh Dandona, SUNY Distinguished Professor, Head of Endocrinology, Diabetes, and Metabolism, State University of New York, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002775; 1987 (Other: Diabetes and Endocrinology Research Foundation)
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; semaglutide; dapagliflozin

STUDY DESIGN:
Intervention Model Description: This will be a two-center, randomized, open-label then double-blind, parallel group, placebo and standard of care controlled prospective study in type 1 diabetes.
Who Masked: Participant, Investigator
Masking Description: This will be a two-center, randomized, open-label then double-blind, parallel group, placebo and standard of care controlled prospective study in type 1 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Standard of care insulin will be used as an active comparator arm for 1/3 of patients (38 patients) for the entire duration of the study.
  Interventions: Drug: Insulin
- Dual Therapy (Experimental): Once a week injection of Semaglutide (a GLP-1 receptor agonist) in addition to standard of care insulin for the first six months in 2/3 of patients (76 patients). Semaglutide is a clear, colorless solution that contains 2 mg of semaglutide in a 1.5 mL (1.34 mg/mL) pre-filled, disposable, single-patient-use pen injector. Semaglutide will be started at the 0.25 mg dose for the first two weeks, then increased to 0.5 mg at week 2, and then yet again increased to 1.0 mg at week 4.
  Interventions: Drug: Insulin; Drug: Semaglutide
- Triple therapy (Experimental): Once a day oral pill (green, plain, diamond shaped film coated 5 mg tablet) of Dapagliflozin (an SGLT-2 inhibitor) added to once a week injection of semaglutide and standard of care insulin in the second 6 months of 1/2 of the dual therapy arm (1/3 of total patients (38 patients)). Dapagliflozin will be started at 5 mg for one week, and then increased to 10 mg for the remainder of the study
  Interventions: Drug: Insulin; Drug: Semaglutide; Drug: Dapagliflozin
- Triple therapy control (Placebo Comparator): Once a day oral pill (green, plain, diamond shaped film coated 5 mg tablet) of the Placebo form of Dapagliflozin added to once a week injection of semaglutide and standard of care insulin in the second 6 months of 1/2 of the dual therapy arm (1/3 of total patients (38 patients)).
  Interventions: Drug: Insulin; Drug: Semaglutide; Drug: Placebo to Dapagliflozin

INTERVENTIONS:
Drug: Insulin — Standard of care insulin for pump or injection and serves as a control
Drug: Semaglutide — Injectable weekly GLP-1RA given as open label experimental drug
  Other Names: Ozempic
  Arms: Dual Therapy; Triple therapy; Triple therapy control
Drug: Dapagliflozin — Oral daily SGLT2 Inhibitor given as experimental drug
  Other Names: Farxigo
  Arms: Triple therapy
Drug: Placebo to Dapagliflozin — Placebo to Dapagliflozin given as a control to the experimental drug
  Arms: Triple therapy control

SUMMARY:
To assess whether the addition of dapagliflozin to semaglutide and insulin (triple therapy) improves glycemic control in patients with type 1 diabetes compared with semaglutide and insulin (dual therapy) and insulin only (standard) treatment.

DETAILED DESCRIPTION:
This will be a 52 week study for type 1 diabetics looking into the effect of semaglutide and dapagliflozin on HbA1c and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes for at least 1 year on staple use of continuous subcutaneous insulin infusion (CSII) or multiple daily (four or more) injections (MDI) of insulin for last 3 months.
2. C-peptide <0.23 nM
3. Minimum dose of insulin in Units/kg at entry: 0.5 U/kg for MDI and 0.4 U/kg for CSII
4. Regularly measuring blood sugars four or more times daily.
5. HbA1c of >7.5%.
6. Well versed in CHO counting*
7. Age 18-70 years.
8. BMI ≥25 kg/m2.

Exclusion Criteria:

1. Type 1 diabetes for less than 12 months, type 2 diabetes, chronic pancreatitis, MODY
2. Previous use of any agent other than insulin for treatment of diabetes in the last 3 months.
3. History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g., emergency room visit and/or hospitalization) within 3 month prior to the screening visit
4. Frequent episodes of severe hypoglycemia as defined by more than one episode requiring medical assistance, emergency care (paramedics or emergency room care), and/or glucagon therapy administered by a third-party individual within 1 month prior to the screening visit
5. Symptoms of poorly controlled diabetes that would preclude participation in this trial
6. Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program
7. History of bariatric surgery or lap-band procedure within 12 months prior to screening
8. History of Addison's disease or chronic adrenal insufficiency
9. History of diabetes insipidus
10. Hepatic disease or cirrhosis with Aspartate Aminotransferase (AST) > 3X Upper limit of normal (ULN) and/or Alanine aminotransferase (ALT) > 3X ULN
11. Serum Total Bilirubin > 2X ULN unless exclusively caused by Gilbert's Syndrome
12. Hemoglobin < 11.0 g/dL (110 g/L) for men; hemoglobin < 10.0 g/dL (100 g/L) for women.
13. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous 3 months or patients with congestive heart failure.
14. ESRD on hemodialysis; and or e-GFR < 60 ml/min/1.73m2
15. HIV or Hepatitis B/C positive status
16. Any other life-threatening, noncardiac disease
17. History of pancreatitis
18. Women who are pregnant or women of childbearing potential who are not using adequate contraception or who are breast feeding
19. Inability to give informed consent
20. History of gastroparesis
21. History of medullary thyroid carcinoma or MEN 2 syndrome
22. History of serious hypersensitivity reaction to these agents
23. Painful gallstones
24. Alcoholism
25. Hypertriglyceridemia (>500 mg/dl)
26. Recurrent genital mycotic infection.
27. Hypovolemic patients or with chronic renal insufficiency.
28. Patients with any malignancy except treated in situ malignancy and basal cell carcinoma of the skin
29. Unexplained hematuria
30. Patients with a history of diabetic retinopathy
31. Use of an investigational agent or therapeutic regimen within 30 days of study
32. Participation in any other concurrent interventional clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c following dapagliflozin | 6 months
  Change in HbA1c at 6 months following dapagliflozin or placebo therapy in addition to combined semaglutide and insulin treatment.

SECONDARY OUTCOMES:
Change in HbA1c with triple therapy | 12 months
  Change in HbA1c from baseline at 12 months in triple therapy group compared to insulin only group.
Change in HbA1c with semaglutide | 6 months
  Change in HbA1c from baseline at 6 months in dual therapy group (insulin and semaglutide) compared to insulin only group.
Assessment of hyperglycemia level 1 | 12 months
  Change in percent Time hyperglycemia Level 1(180-250mg/dl) as assessed by CGM
Assessment of hyperglycemia level 2 | 12 months
  Change in percent Time in hyperglycemia Level 2 ( >250mg/dl) as assessed by CGM
Assessment of hypoglycemia | 12 months
  Change in percent Time in hypoglycemia Level 1 (54-70mg/dl) as assessed by CGM
Assessment of percent time glucose in range | 12 months
  Change in percent Time in Range (70- 180 mg/dl) as assessed by CGM
Fructosamine indices | 12 months
  Assessment of fructosamine
Weekly fasting glucose indices | 12 months
  Assessment of change of weekly fasting glucose
Insulin requirement indices | 12 months
  Assessment of the change in insulin requirement
body weight assessment following dapagliflozin | 6 months
  Change in body weight at 6 months between dapagliflozin and placebo groups.
body weight assessment following semaglutide | 6 months
  Change in body weight at 6 months following starting semaglutide compared to standard of care (SOC) group.
body weight assessment following triple therapy | 12 months
  Change in body weight as assessed at 12 months on dapagliflozin and semaglutide compared to SOC therapy.
Systolic Blood pressure assessment after triple therapy | 12 months
  Anti-hypertensive effects including change in systolic BP on dapagliflozin and semaglutide compared to SOC therapy.
Diastolic Blood pressure assessment | 12 months
  Anti-hypertensive effects including change in diastolic BP on dapagliflozin and semaglutide compared to SOC therapy.
Blood pressure medication use | 12 months
  Anti-hypertensive effects including change in numbers of BP medications required in patients dapagliflozin and semaglutide compared to SOC therapy.
Level 2 hypoglycemia assessment | 12 months
  Differences in rates of hypoglycemic events Level 2 (<54mg/dl) between triple therapy and in standard therapy arm.
Severe (level 3) hypoglycemia assessment | 12 months
  Differences in rates of hypoglycemic events Level 3 (<54mg/dl) characterized by altered mental and/or physical status requiring assistance) between triple therapy and in standard therapy arm.
Level 1 hyperglycemia assessment | 12 months
  Differences in rates of Level 1 hyperglycemia (glucose levels >180mg/dl and <250mg dl) between triple therapy and in standard therapy arm.
Level 2 hyperglycemia assessment | 12 months
  Differences in rates of Level 2 hyperglycemia (glucose levels <250mg dl) between triple therapy and in standard therapy arm.
serum ketones assessment | 12 months
  Differences in rates of diabetic ketoacidosis defined as elevated serum ketones (greater than the upper limit of the normal range) in investigative arms.
Urinary ketones assessment | 12 months
  Differences in rates of diabetic ketoacidosis defined as elevated urine ketones (greater than the upper limit of the normal range) in investigative arms.
Diabetic ketoacidosis assessment | 12 months
  Differences in rates of diabetic ketoacidosis defined as Blood pH <7.3 in investigative arms.

CONTACTS AND LOCATIONS:
Overall Officials: Husam Ghanim, PhD, Study Director — State University of NY at Buffalo
Locations (1):
- Diabetes and Endocrinology Research Center of WNY, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT03899402/Prot_000.pdf